CLINICAL TRIAL: NCT07113249
Title: The Effects of Foam Rolling During the Warm-Up Phase on Range of Motion, Ankle Stability and Leaping Performance in Young Elite Rhythmic Gymnasts
Brief Title: The Effects of Foam Rolling on Ankle Dorsiflexion, Ankle Stability, and Athletic Performance in Rhythmic Gymnasts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Giacomo Belmonte, Dr., University of Palermo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 62141-2025-1
Record Dates: First submitted 2025-08-02; First posted 2025-08-08 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-07

CONDITIONS: Athletes
Keywords: Rhythmic Gymnasts; Performance; Injury Prevention

STUDY DESIGN:
Intervention Model Description: Experimental Group (EG) and Control Group (CG)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Foam Rolling (FR) (Experimental): Three sets, each lasting 60 seconds, with a 30-second break between sets for two times for week. During each FR session, a complete sequential movement was always performed, starting from the gastrocnemius muscles and ending with the soleus. A metronome was set to play one complete repetition every 2 seconds to establish the speed of execution.
  Interventions: Other: Foam Rolling (FR)
- Control Group (CG) (No Intervention)

INTERVENTIONS:
Other: Foam Rolling (FR) — For the FR, participants were asked to place the roller behind their leg. Three sets, each lasting 60 seconds, with a 30-second break between sets, were performed, for a total of 90 rolls per set.
  Arms: Experimental: Foam Rolling (FR)

SUMMARY:
Rhythmic Gymnastics is an Olympic discipline featuring individual or team competition. Regardless of the type of competition, athletes undergo rigorous training focused on enhancing their coordination, joint range of motion, and jump height. Each rhythmic gymnast voluntarily underwent testing at their own gym after reading and signing the informed consent document. During the first session, general information was collected on all participants (age, weight, and height), followed by an assessment of athletic performance and joint mobility parameters. For the jump performance parameters, the Counter Movement Jump test (CMJ) was used through an optical detecting system. An inertial sensor was used to measure joint mobility, while a pressure platform was used to measure ankle stability, using a single-leg jump protocol. Subsequently, participants were randomly divided into two groups: an experimental group (EG) and a control group (CG). The EG performed three sets, each lasting 60 seconds, with a 30-second break between sets for two times for week for 3 weeks. During each FR session, a complete sequential movement was always performed, starting from the gastrocnemius muscles and ending with the soleus muscle. At the end of the three weeks, all measurements were repeated.

ELIGIBILITY:
Inclusion Criteria:

* Active participation in competitive training programs (at least 10 hours per week), at least one year of experience in competitions organized by the Italian Gymnastics Federation, and no recent injuries.

Exclusion Criteria:

* Presence of current or not fully recovered injuries to the ankle or foot, and irregular participation in training sessions within the four weeks preceding the study.

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Counter Movement Jump (CMJ) | At the beginning of enrollment ( Baseline, T0) and the end of the 3-week treatment (T1)
  Initially, the athlete stands upright on a flat surface or force platform, feet shoulder-width apart, hands on hips (to eliminate arm swing). Without a pause, the athlete performs a quick downward movement (countermovement) by bending the knees and hips, then immediately jumps vertically as high as possible. The athlete lands in an upright position on the same spot, trying to absorb the impact with knees slightly bent. Jump height and flight time is recorded using an optical system, Optojump™ system(Microgate, Bolzano, Italy) connected to a personal computer with dedicated software(OptojumpTM Next software). The system consists of two optical bars, a receiver and a transmitter, positioned 1m apart. The bars identify ground contact time(with a precision of 1ms) and then convert non-contact time into cm. Based on recommendations on optimal jump height (20 to 60cm).
Ankle Dorsiflexion ROM | At the beginning of enrollment ( Baseline, T0) and the end of the 3-week treatment (T1)
  Each participant was fitted with an inertial sensor (Beyond Inertial, Motusech, Roma, Itay) in the center of the foot, using an elastic band supplied with the sensor. The starting position was standardized with the subjects sitting on a medical bed with the popliteal cord attached to the edge of the bed, forming a 90° angle. The position of the foot, on the other hand, was placed in a neutral position using a laser level. Subsequently, the dorsal flexion movement was performed.
Ankle Stability | At the beginning of enrollment ( Baseline, T0) and the end of the 3-week treatment (T1)
  Ankle stability was assessed using a functional monopodalic protocol, which involved four jumps on one foot: two per leg, both frontally and laterally. These jumps were performed by stepping over an adjustable obstacle set at 70% of the maximum height reached on a pressure platform (SensorMedica freeMed 40×40, Guidonia Montecelio, Italy). The platform has an active sensory surface of 40×40 cm with a thickness of only 8 mm and a low weight of approximately 4 kg. Inside, there are resistive sensors coated in 24K gold on conductive rubber, with a density of approximately 10,000 sensors/m².The acquisition frequency is high, up to 400 Hz, allowing for detailed dynamic analysis, and the sensors have a life cycle of over 1,000,000 cycles of use

CONTACTS AND LOCATIONS:
Locations (1):
- University of Palermo, Palermo, Italy, Italy

REFERENCES:
- [Derived] Belmonte G, Patti A, Di Mitri IR, Gervasi M, Formiglio E, Fernandez-Pena E, Thomas E, Bianco A. Effects of a 3-week foam rolling warm-up intervention on ankle dorsiflexion measurements and jumping performance in young rhythmic gymnasts. BMC Sports Sci Med Rehabil. 2026 Feb 10. doi: 10.1186/s13102-026-01575-2. Online ahead of print. PMID 41664208